CLINICAL TRIAL: NCT02840227
Title: The Effect of Combined General/Regional Anesthesia on Cancer Recurrence in Patients Having Lung Cancer Resections
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Shanghai Chest Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 091051
Record Dates: First submitted 2016-06-20; First posted 2016-07-21 (Estimated); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Cancer; General anesthesia; Epidural anesthesia
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — Anesthesia, General; Anesthesia, Epidural

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Combined general/epidural anesthesia (Experimental): Combined general/epidural anesthesia and analgesia. General anesthesia may include propofol, isoflurane, sevoflurane, and other drugs. Epidural anesthesia will include bupivacaine and other local anesthetics.
  Interventions: Procedure: Combined general/epidural anesthesia
- General anesthesia with opioid analgesia (Experimental): General anesthesia with routine drugs and intravenous PCA opioid analgesia. General anesthesia may include propofol, isoflurane, sevoflurane, and other drugs.
  Interventions: Procedure: General anesthesia with opioid analgesia

INTERVENTIONS:
Procedure: General anesthesia with opioid analgesia — General anesthesia with routine drugs and intravenous patient controlled opioid analgesia. General anesthesia may include propofol, isoflurane, sevoflurane, and other drugs.
  Arms: General anesthesia with opioid analgesia
Procedure: Combined general/epidural anesthesia — Combined general/epidural anesthesia and analgesia. General anesthesia may include propofol, isoflurane, sevoflurane, and other drugs. Epidural anesthesia will include bupivacaine and other local anesthetics.
  Arms: Combined general/epidural anesthesia

SUMMARY:
The primary hypothesis is that disease-free survival is improved in patients undergoing resection for tumor thought to be stage I-III primary non-small cell lung cancer in patients with combined general-epidural anesthesia & analgesia as compared to patients receiving general anesthesia and postoperative patient-controlled opioid analgesia. Patients having surgery for resection of potentially curable lung cancer will be randomized to combined general and epidural anesthesia or general anesthesia with opioid analgesia. The primary outcome will be disease-free survival.

DETAILED DESCRIPTION:
Surgery is the primary treatment of lung cancer, but surgery releases tumor cells into the systemic circulation. Whether this minimal residual disease results in clinical metastases is a function of host defense. At least three perioperative factors shift the balance toward initiation and progression of minimal residual disease.

1. Surgery per se depresses cell-mediated immunity, reduces concentrations of tumor-related anti-angiogenic factors (e.g., angiostatin and endostatin), and increases concentrations of pro-angiogenic factors such as VEGF.
2. Anesthesia impairs numerous immune functions, including neutrophil, macrophages, dendritic cells, T-cell, and NK-cell functions.
3. Opioid analgesics inhibit both cellular and humoral immune function in humans, and promote tumor growth in rodents.

The primary hypothesis is that disease-free survival is improved in patients undergoing resection for tumor thought to be stage I-III primary non-small cell lung cancer in patients with combined general-epidural anesthesia & analgesia as compared to patients receiving general anesthesia and postoperative patient-controlled opioid analgesia. Patients having surgery for resection of potentially curable lung cancer will be randomized to combined general and epidural anesthesia or general anesthesia with opioid analgesia. The primary outcome will be disease-free survival.

The effect of combined epidural/general anesthesia versus general anesthesia with opioid analgesia on the primary outcome of disease-free survival (time to the earlier or recurrence or death from any cause) will be assessed uni-variably with Kaplan-Meier analyses and multivariably (primary analysis) with a Cox proportional hazards regression model adjusting for known risk factors for recurrence, including tumor stage, size of tumor, age, sex, receipt of chemotherapy before or after surgery, and clinical site. As usual for this type of analysis, stopping criteria will be based on number of outcome events rather than enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Tumor thought to be primary non-small cell lung cancer (stage 1-3) as determined according to the IASLC Lung Cancer Staging Project[ref];
2. Scheduled for potentially curative tumor resection;
3. Written informed consent, including willingness to be randomized to epidural anesthesia/analgesia plus general anesthesia or to general anesthesia and postoperative opioid analgesia;
4. ASA physical status 1-3.

Exclusion Criteria:

1. Any contraindication to epidural anesthesia, (including coagulopathy, abnormal anatomy).
2. Any contraindication to midazolam, propofol, sevoflurane, fentanyl, morphine, or hydromorphone.
3. Age <18 or >85 years old.
4. Other cancer not believed by the attending surgeon to be in long-term remission.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Cancer-free survival | 3 years or as available
  Patients who remain alive without known lung cancer recurrence

SECONDARY OUTCOMES:
Pain intensity | 2 days
  Time-weighted average pain scores over initial two days of hospitalization.
SF-12 Health Survey | 6, 12, 24, and 36 months
McGill Pain Questionnaire | 6, 12, 24, and 36 months
Neuropathic Pain Questionnaire | 6, 12, 24, and 36 months
Opioid use | 2 days
  Total opioid use

CONTACTS AND LOCATIONS:
Overall Officials: Daniel I Sessler, MD, Study Chair — The Cleveland Clinic
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No